CLINICAL TRIAL: NCT01770613
Title: A PHASE IIa, DOUBLE-BLINDED, MULTI-CENTER, RANDOMIZED STUDY TO ASSESS THE SAFETY,TOLERABILITY, AND PRELIMINARY EFFICACY OF A SINGLE INTRAVENOUS DOSE OF ALLOGENEIC MESENCHYMAL BONE MARROW CELLS TO SUBJECTS WITH ST SEGMENT ELEVATION MYOCARDIAL INFARCTION (STEMI)
Brief Title: A Study of Allogeneic Mesenchymal Bone Marrow Cells in Subjects With ST Segment Elevation Myocardial Infarction (STEMI)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate business decision, may consider different subject population
Sponsor: Stemedica Cell Technologies, Inc. (Industry)
Collaborators: CardioCell LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEM 103-M-STEMI
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: ST Segment Elevation Myocardial Infarction (STEMI); Allogeneic Mesenchymal Bone Marrow Cells
Keywords: Adult; Allogeneic; Stem; Cells; Myocardial; Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cells (Experimental): ALLOGENEIC MESENCHYMAL BONE MARROW CELLS
  Interventions: Biological: Stem cells
- Control (Placebo Comparator): Lactated Ringer's Solution
  Interventions: Biological: Stem cells

INTERVENTIONS:
Biological: Stem cells — Allogeneic mesenchymal stem cells

SUMMARY:
The purpose of this study is to assess the safety and tolerability of human allogeneic mesenchymal bone marrow cells (aMBMC) administered intravenously to subjects with ST Segment Elevation Myocardial Infarction (STEMI).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains a leading cause of morbidity and mortality despite continuing advances in various treatment options. In developed countries, ischemic heart disease causes more than 50% of all cardiovascular deaths. It is estimated that one in three or approximately 80 million American adults have one or more types of CVD, with approximately 38.1 million of those estimated to be 60 years of age or older. The data was extrapolated to the United States population in 2006 from National Health and Nutrition Examination Survey (NHANES) 2005-2006 data.

Mortality data show CVD as the underlying cause of death (including congenital cardiovascular defects) accounting for 35.3% (864,480) of all 2,448,017 deaths in 2005, or one of every 2.8 deaths in the United States. CVD total deaths (1,372,000 deaths in 2005) accounted for about 56% of all deaths in 2005. Nearly 2,400 Americans die of CVD each day, an average of one death every 30 seconds. CVD claims about as many lives each year as cancer, chronic lower respiratory diseases, accidents, and diabetes mellitus combined (NCHS).

Stem cell transplantation has the potential to repair and improve cardiac function, thus helping to significantly decrease morbidity and mortality rates. Preclinical data from a variety of animal studies demonstrated the capacity for skeletal myoblasts to engraft, form myotubules, and enhance cardiac function after transplantation into infarcted myocardium. The underlying sequela of the post infarcted left ventricle often includes massive damage to the cardiomyocyte. The left ventricle remodeling (dilation) and dysfunction is thought to be irreversible. The development of treatments that will regenerate its musculature and vascular components is now considered a main therapeutic challenge. Preliminary human studies focusing on subjects with ischemic heart disease have demonstrated successful myoblast transplantation into the post infarction scar. Another study demonstrated the benefits of stem cell therapy on ventricular function and profusion. Dib et. al., demonstrated the survival, feasibility, and safety of autologous myoblast transplantation and suggests that stem cell transplantation offers a potential therapeutic treatment for end-stage heart disease.

Allogeneic mesenchymal stem cells have been used in a number of clinical trials for different indications. These clinical trials demonstrated the safety of allogeneic mesenchymal stem cell treatment. Allogenic mesenchymal bone marrow cells can be isolated from bone marrow. They are the primary cells used in tissue engineering expressing multiple cell types. Tissue engineering is very promising, generating hope that reconstruction of organs and repair diseased and damaged tissue may be possible.

There are two major types of aMBMC, hematopoetic (mononuclear) and stromal MSCs. Stromal MBMC, the cell type to be used in this study, proved to be more effective in reestablishing profusion as they secreted additional cytokine factors associated with angiogenesis. The multilineage potential of stromal MSCs, their ability to elude detection by the host immune system and even down regulate T-cell response allows for allogeneic multiple stem cell therapeutic use.

Occlusion of the left main or left anterior descending artery causes irreversible injury to the cardiomyocytes in as little as 20 minutes. The goal of therapy in ischemic cardiomyopathy is to limit damage in the following areas:

* Limit infarct size
* Prevent reperfusion injury
* Prevent excessive fibrosis
* Reestablish function of hibernating cardiomyocytes in peripheral zone area.
* Reestablish angiogenesis/vasculogenesis
* Preserve wall motion (prevent arrhythmia and functional contractile deterioration)
* Prevent post infarct ventricular remodeling and left ventricular dilation It is well accepted that dilated cardiomyopathy mortality rates are 50% within 5 years of diagnosis. If we can preserve and restore cardiac function as measured by ejection fraction, preserving left ventricular integrity would increase subject quality of life as well as longevity.

An IV study administering adult allogeneic mesenchymal stem cells (MSC) to 53 subjects following AMI showed excellent safety, reduction in arrhythmias, improvement in functional status and increased ejection fraction. The availability of "off the shelf" allogeneic stem cells will allow for an easily adjustable dose (getting enough cells in the autologous model is often a problem) for each individual subject. The ease of IV administration will make stem cell therapy more cost effective and safer to administer than the current catheter models. This study protocol will expand on the safety and efficacy of aMBMC in subjects suffering from ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-85 years of age.
2. First ST Segment Elevation Myocardial Infarction (STEMI) of ischemic etiology affecting the left ventricle within 7 days of study enrollment. Myocardial infarction is defined as ECG evidence of clinically significant ST-segment elevation (>1mm [0.1 mV] in at least 2 contiguous precordial leads or in at least 2 adjacent limb leads).
3. Subject had successful revascularization within 12 hours of symptoms as evidenced by residual stenosis < 30% and TIMI antegrade flow II or III in the culprit vessel. Revascularization may include one of the following:

   * PCI angioplasty/stenting placement
   * Thrombolytic therapy
4. LVEF ≤45% as determined by 16-lead quantitative 2D echocardiography more than 24 hours after revascularization.
5. Life expectancy greater than 12 months.
6. Ability to understand and provide signed informed consent, or have a designated legal guardian or spouse legally able and willing to make such decisions on the subject's behalf.
7. Reasonable expectation that subject will receive standard post myocardial infarction care, unless contraindicated, including medications:

   • Anticoagulation (e.g. aspirin, clopidogrel, ticlopidine, prasugrel, etc.), beta-blockers, ace inhibitors, and statin agents, as tolerated.
8. Attend all scheduled safety follow-up visits.

Exclusion Criteria:

1. Hemodynamic instability as demonstrated by any of the following:

   1. Requirement of intra-aortic balloon pump of left ventricular assist device.
   2. Need for inotropic support (e.g. dopamine and/or dobutamine) for more than 36 hours for the maintenance of mean arterial blood pressure ≥60 mmHg.
2. History of cancer within the past 5 years, with the exception of localized basal or squamous cell carcinoma.
3. Clinically-significant hematologic, hepatic, or renal impairment within 24 hours of study procedure as determined by screening clinical laboratory tests. Severe chronic anemia or hematocrit ≤24%. Liver function tests (total bilirubin at 3 times upper limit of normal, or creatinine level ≥3mg/dL).
4. Presence of any other clinically-significant medical condition, psychiatric condition, or laboratory abnormality, that in the judgment of the Investigator or Sponsor for which participation in the study would pose a safety risk to the subject.
5. Participation in another study with an investigational drug or device within 3 months prior to stem cell administration.
6. History within the past year of drug or alcohol abuse.
7. Females known to be pregnant, lactating or having a positive pregnancy test (will be tested during screening) or planning to become pregnant during the study.
8. Inability to comply with the conditions of the protocol.
9. Presence of a transplanted tissue or organ or left ventricular assist device (LVAD) (or the expectation of the same within the next 12 months).
10. Planned Automatic Implantable Cardiac Defibrillator (AICD) or CRT within the next 12 months.
11. Need for chronic intermittent inotropic therapy.
12. Active myocarditis or early postpartum cardiomyopathy (within the first twelve months of delivery).
13. Systemic corticosteroids, cytostatics, immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), and DNA depleting or cytotoxic drugs taken within four weeks prior to study stem cell administration.
14. Porphyria.
15. Allergy to sodium citrate or any "caine" type of local anesthetic.
16. Subject scheduled for hospice care.
17. Clinically relevant abnormal findings in the clinical history, physical examination, ECG (e.g. life threatening arrhythmias, including QTc interval of ≥550 ms) or laboratory tests at the screening assessment that would interfere with the objectives of the study or that would, in the Investigator's opinion, preclude safe completion of the study.
18. Abnormal findings could include: known HIV infection or other immunodeficiency state, chronic active viral infection (such as hepatitis B or C), acute systemic infections (defined as subjects undergoing treatment with antibiotics), gastrointestinal tract bleeding, or any severe or acute concomitant illness or injury.
19. Any other medical, social, or geographical factor that would make it unlikely that the subject could comply with study procedures (e.g., alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location, or a history of noncompliance).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of aMBMC intravenous administration during the twelve month study period as determined by major adverse events MACE endpoint. | 12 months

SECONDARY OUTCOMES:
The change from baseline on physical exam conducted at day 14 and at 1, 3, 6 and 12 months post-administration, as available: | 12 months
• LV end diastolic volume | 12 months
• LV end systolic volume | 12 months
• Infarct size measured by MRI, with and without contrast (only for patients eligible for MRI) | 12 months
• Global Left Ventricular Ejection Fraction (measured by echocardiography) | 12 months
• SF-36 Health Assessment | 12 months
• Incidence of Ventricular Arrhythmias requiring intervention at 1 and 3 months post-administration | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Dib, MD, MSc, FACC, Principal Investigator — Mercy Gilbert Medical Center, Dignity Health
Locations (2):
- United States (2):
  - Mercy Gilbert and Chandler Medical Center, Gilbert, Arizona
  - Emory University Hospital, Atlanta, Georgia